CLINICAL TRIAL: NCT04259372
Title: Analysis of T Cell Metabolism and Immune Phenotype During the Course of Acute Myeloid Leukemia
Brief Title: Analysis of T Cell Metabolism in Acute Myeloid Leukemia Patients
Status: Completed | Type: Observational
Sponsor: University of Freiburg (Other)
Responsible Party: Principal Investigator, Robert Zeiser, Director of the Division of Tumor Immunology, University of Freiburg
Other Study IDs: Tmet_AML
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Primary Diagnosis: Analysis of patient blood at primary diagnosis of AML
- Relapse: Analysis of patient blood at time point of relapse after allo-HCT
- Remission: Analysis of patient blood during remission after allo-HCT

SUMMARY:
The objective of this study was to analyze the T cell metabolism and immune phenotype in AML patients during the course of the disease before and after allo-HCT.

DETAILED DESCRIPTION:
Patients who experience relapse of acute myeloid leukemia (AML) after allogeneic hematopoietic cell transplantation (allo-HCT) have a dismal prognosis. Infusion of donor T cells can induce graft-versus-leukemia (GVL) effects, indicating the importance of intact T cell function for leukemia control. Recent studies have shown the importance of metabolic fitness for an effective T cell response.

In this study we have analyzed the T cell metabolism and immune phenotype in AML patients at different time points before and after allo-HCT.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of AML
* age ≥ 18 years
* peripheral blood sample available
* written informed consent
* ability to understand the nature of the study and the study related procedures and to comply with them

Exclusion Criteria:

* age < 18 years
* lack of informed consent
* patients that cannot be classified in one of the 3 groups

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with acute myeloid leukemia at primary diagnosis, at relapse after allo-HCT or in remission after allo-HCT.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
T cell metabolism | 4 years
  Extracellular acidification rate (ECAR) and oxygen consumption rate (OCR) determined by live-cell metabolic assay using the Seahorse Analyzer
T cell phenotype | 4 years
  T cell cytokine and effector molecule production

SECONDARY OUTCOMES:
Metabolite abundance in serum | 4 years
  Serum metabolites as measured by mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zeiser, Prof. Dr., Principal Investigator — Medical Center University of Freiburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buck MD, O'Sullivan D, Klein Geltink RI, Curtis JD, Chang CH, Sanin DE, Qiu J, Kretz O, Braas D, van der Windt GJ, Chen Q, Huang SC, O'Neill CM, Edelson BT, Pearce EJ, Sesaki H, Huber TB, Rambold AS, Pearce EL. Mitochondrial Dynamics Controls T Cell Fate through Metabolic Programming. Cell. 2016 Jun 30;166(1):63-76. doi: 10.1016/j.cell.2016.05.035. Epub 2016 Jun 9. PMID 27293185
- [Background] Chang CH, Qiu J, O'Sullivan D, Buck MD, Noguchi T, Curtis JD, Chen Q, Gindin M, Gubin MM, van der Windt GJ, Tonc E, Schreiber RD, Pearce EJ, Pearce EL. Metabolic Competition in the Tumor Microenvironment Is a Driver of Cancer Progression. Cell. 2015 Sep 10;162(6):1229-41. doi: 10.1016/j.cell.2015.08.016. Epub 2015 Aug 27. PMID 26321679
- [Background] Schmid C, Labopin M, Nagler A, Bornhauser M, Finke J, Fassas A, Volin L, Gurman G, Maertens J, Bordigoni P, Holler E, Ehninger G, Polge E, Gorin NC, Kolb HJ, Rocha V; EBMT Acute Leukemia Working Party. Donor lymphocyte infusion in the treatment of first hematological relapse after allogeneic stem-cell transplantation in adults with acute myeloid leukemia: a retrospective risk factors analysis and comparison with other strategies by the EBMT Acute Leukemia Working Party. J Clin Oncol. 2007 Nov 1;25(31):4938-45. doi: 10.1200/JCO.2007.11.6053. Epub 2007 Oct 1. PMID 17909197